CLINICAL TRIAL: NCT04049409
Title: A Randomized, Double-blinded, Controlled, Single Dosing Phase I Study to Investigate The Pharmacokinetic, Safety and Immunogenicity Characteristics of CMAB809 and Herceptin in Healthy Male Subjects
Brief Title: Pharmacokinetic, Safety and Immunogenicity Study of CMAB809 and Herceptin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taizhou Mabtech Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: CMAB809HV-I
Record Dates: First submitted 2019-07-16; First posted 2019-08-08 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMAB809 (Experimental)
  Interventions: Drug: CMAB809
- Trastuzumab (Active Comparator)
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: CMAB809 — CMAB809 will be administered by IV infusion at a single dose of 6mg/kg.
  Arms: CMAB809
Drug: Trastuzumab — Trastuzumab will be administered by IV infusion at a single dose of 6mg/kg.
  Arms: Trastuzumab

SUMMARY:
This is a randomized, double-blinded, controlled Phase I study of CMAB809 administered by intravenous infusion. This study will characterize the pharmacokinetic, safety and immunogenicity of CMAB809 versus Trastuzumab(Herceptin) in healthy male subjects after a single dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, age ranged 18 to 45 years (both inclusive)
* A subject with body weight be equal or greater than 50 kg (inclusive) and body mass index (BMI) between 19 and 26 kg/m2 (both inclusive)
* Findings within the range of clinical acceptability in medical history and physical examination, and laboratory results within the laboratory reference ranges for the relevant laboratory tests (unless the investigator considers the deviation to be irrelevant for the purpose of the study)
* Left ventricular ejection fraction (LVEF) within the normal range by echocardiogram (ECHO) at 2 weeks prior to randomization
* The subjects have the ability to understand the full characteristics and objectives of the study, including the possible risks and side effects of the study; Moreover, the subjects can communicate well with researchers and complete the research according to the regulations
* Subjects must voluntarily sign ICF prior to the study

Exclusion Criteria:

* Any clinical signs and symptoms (including blood pressure, pulse, and electrocardiogram) found during medical examination; And those who underwent surgery within 4 weeks before screening; Or plans to operate during the trial period
* Diagnosed with any clinical history of serious illness or any other disease or physiological conditions which can interfere with the test results
* Prescription or over-the-counter drugs with a long half-life (greater than 24h) within 1 month prior to administration. Take any other medication that the investigator considers may affect the subject's enrollment within 2 weeks prior to administration. A subject who has participated in any other clinical trial within 3 months before the study drug administration
* Have used or are using biological products such as monoclonal antibodies or fusion proteins
* Patients who have or have had chronic hepatitis b, c, syphilis or HIV infection, or who have tested positive for the above infection were deemed unsuitable to participate in this study
* Those who had been vaccinated within 30 days prior to screening or who needed to be vaccinated between screening and the end of the trial
* Drug abusers, or those who used soft drugs (e.g., marijuana) 3 months before screening, or took hard drugs (e.g., cocaine, phenyclohexidine, etc.) 1 year before the test, or drank excessive amounts of tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup =250ml) every day, or those who showed positive urine drug screening
* Blood donation (containing component blood) or lost more than 400 mL of blood within 3 months before screening, or blood transfusion; Blood donation (containing component blood) or blood loss of more than 200 mL within 1 month before screening
* Related allergies (including allergy to any mouse\human protein or immunoglobulin products, rubber or latex)
* Those who smoked more than 10 cigarettes per day within 6 months before screening; And those who could not quit during the study period
* Alcoholics (who drink more than 14 standard units per week), or who have positive result in breath-test of alcohol
* Vigorous activity for 72h before drug administration; and cannot be avoided within 7 days after drug administration
* Unable to accept clinical trial center diet
* Fertile men who were unwilling to use highly effective contraceptives during the trial and for five months after administration
* The investigator judges the subject not eligible for the study after reviewing clinical laboratory results or other reasons

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve [AUC] | pre-dose, hour1.5, hour3, hour8, hour24, hour48, hour96, hour168, hour336, hour504, hour672, hour1008, hour1344, hour1680 post-dose
  Area under the concentration-time curve [AUC] from 0 to the last time point selected of CMAB809

SECONDARY OUTCOMES:
Cmax | pre-dose, hour1.5, hour3, hour8, hour24, hour48, hour96, hour168, hour336, hour504, hour672, hour1008, hour1344, hour1680 post-dose
  Maximum Serum Concentration(Cmax) of CMAB809
AUC0-∞ | pre-dose, hour1.5, hour3, hour8, hour24, hour48, hour96, hour168, hour336, hour504, hour672, hour1008, hour1344, hour1680 post-dose
  Area under the concentration-time curve from 0 to inf(AUC0-∞) of CMAB809
Tmax | pre-dose, hour1.5, hour3, hour8, hour24, hour48, hour96, hour168, hour336, hour504, hour672, hour1008, hour1344, hour1680 post-dose
  The time of maximum blood concentration after administration(Tmax) of CMAB809
CL | pre-dose, hour1.5, hour3, hour8, hour24, hour48, hour96, hour168, hour336, hour504, hour672, hour1008, hour1344, hour1680 post-dose
  Total clearance after bioavailability correction(CL) of CMAB809
T1/2 | pre-dose, hour1.5, hour3, hour8, hour24, hour48, hour96, hour168, hour336, hour504, hour672, hour1008, hour1344, hour1680 post-dose
  Half-life(T1/2) of CMAB809
Vd | pre-dose, hour1.5, hour3, hour8, hour24, hour48, hour96, hour168, hour336, hour504, hour672, hour1008, hour1344, hour1680 post-dose
  Apparent volume of distribution corrected for bioavailability(Vd) of CMAB809

OTHER OUTCOMES:
Percentage of participants with Adverse Events | Up to 71 days after administration
  Percentage of participants with Adverse Events (AEs) according to National Cancer Institute Common Terminology Criteria for AEs, Version 5.0(NCI CTCAE V5.0) Common Terminology Criteria for AEs, Version 5.0 (NCI CTCAE V5.0)
anti-drug antibodies(ADA) | pre-dose, week3, week5 and week11 post-dose
  The number of subjects will be summarized
anti-drug antibodies(ADA) | pre-dose, week3, week5 and week11 post-dose
  The percentage of subjects will be summarized
Neutralization antibodies(Nab) | pre-dose, week3, week5 and week11 post-dose
  The number of subjects will be summarized
Neutralization antibodies(Nab) | pre-dose, week3, week5 and week11 post-dose
  The percentage of subjects will be summarized

CONTACTS AND LOCATIONS:
Overall Officials: Jingying Jia, MSC, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China